CLINICAL TRIAL: NCT04985149
Title: Evaluation of the Sural Nerve With Ultrasonography and Electromyography in Patients With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Aysun Ozlu, Principal Investigator, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-02/02
Record Dates: First submitted 2021-07-06; First posted 2021-08-02 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-06

CONDITIONS: Fibromyalgia
Keywords: Pain; fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup 1; participants with fibromyalgia (Other): Participants with fibromyalgia
  Interventions: Other: Electromyographic measurement:; Other: Ultrasonographic measurement:
- Grup 2: patients without fibromyalgia (Other): Patients without fibromyalgia
  Interventions: Other: Electromyographic measurement:; Other: Ultrasonographic measurement:

INTERVENTIONS:
Other: Electromyographic measurement: — Nerve conduction studies; assesses nerve function and includes motor, sensory, and mixed nerve tests.
  Micromed (Italy 2020) EMG device will be used in the electrophysiological examination. Sensory and motor conduction studies will be performed in the lower and upper extremities by paying attention to the extremity temperatures of the cases.
  Nerve conduction studies will be performed by another physician who is unaware of the diagnosis of the patients. Bilateral lower extremity sural sensory responses of the patients will be taken.
  In the antidromic method in sural nerve conduction examination, the bipolar superficial electrode is placed behind the lateral malleolus; stimulation will be made with bipolar surface electrodes 12-15 cm proximal to the recording site. Initial latency should be < 3.8 ms, amplitude > 10 Mv, and conduction velocity > 36 m/sec in sensory response of the sural nerve.
Other: Ultrasonographic measurement: — Sural nerve ultrasonography (US) will be performed by another clinician (Merve Akdeniz leblebicier) who is experienced in musculoskeletal ultrasonography and unaware of clinical evaluation, using a 6-18 Mhz linear probe. (Mindray -UMT 200, United States) Both sural nerve joints of the patients will be evaluated. The patient will lie on the stretcher in the prone position, the ankle will be out of the bed. The 14 cm above the malleolus will be marked as the main line, the nerve will be detected in the lateral of the tendon of the gastrocnemius muscle and the proximal of the saphenous vein. Nerve diameter measurement will be measured 3 times in mm2 and the average will be taken. Then, possible inflammatory pathologies will be ruled out by providing clinical confirmation using the Doppler mode (11).

SUMMARY:
By evaluating the ultrasonographic and electromyographic measurements of the sural nerve in patients with and without a diagnosis of fibromyalgia; to determine the relationship of these measures to each other and to the FIQ, neuropathic pain questionnaire-Clinical, single-blind, prospective, controlled study.

DETAILED DESCRIPTION:
In this study; the investigators will compare the results by evaluating the ultrasonographic and electromyographic measurements of the sural nerve between the groups and determine correlation of these results to each other and to the FIQ, neuropathic pain questionnaire in both groups.

Where the research will be conducted:

Kütahya Health Science Univercity Department of Physical Medicine and Rehabilitation Department The planned date range of the research: August 15 th 2021- December 2021 In the research; the investigators will include 55 participants who were diagnosed with fibromyalgia and 55 participants who were not diagnosed with fibromyalgia meeting the inclusion and exclusion criteria in Kütahya Health Sciences University Evliya Çelebi Training and Research Hospital between August 15 th 2021- December 2021, Participants without fibromiyalgia were planned as control group. All Participants will be asked about their age, gender, marital status, occupation, chronic diseases and previous surgeries, height-weight, smoking-alcohol use, when the diagnosis of fibromyalgia was and the drugs they used and also past operations.

This study is a single-blind, prospective study. The sural nerve electromyographic study, ultrasonographic measurement of the sural nerve, Fibromyalgia Impact Questionnaire and Neuropathic Pain Questionnaire will be applied by obtaining the consent of both groups.

Sample Selection: Computerized rondomized sample selection will be made. Statistical method to be used: The data to be obtained as a result of the study will be analyzed with the SPSS 20.0 statistical package program. Descriptive information will be given by calculating mean, frequency distributions, minimum, maximum, standard deviation, and percentage values. Whether there is a significant difference between the two groups by looking at the means will be evaluated with the independent student t test. The incidence of abnormal tests in EMG and US findings, and comparison of tests and examination findings will be made with the ANOVA test. Continuous variables will be given as mean±standard deviation and categorical variables as frequency and percentage. P values less than 0.05 will be considered statistically significant and the results will be evaluated.

In the Power analysis and sampling calculation made for our study, a total of 100 people can be included in the study by taking the alpha value (p) 0.05 with 95% power. (50 controls / 50 cases). The calculation was made with the G*Power 3.1.9.4 program.

Grup 1; Participants with fibromyalgia Grup 2: Participants without fibromyalgia (Control group)

Interventions:

Sural Nerve Electromyographic measurement:

Nerve conduction studies; assesses nerve function and includes the motor, sensory, and mixed nerve tests.Micromed (Italy 2020) EMG device will be used in the electrophysiological examination. Sensory and motor conduction studies will be performed in the lower and upper extremities by paying attention to the extreme temperatures of the cases. Nerve conduction studies will be performed by another physician who is unaware of the diagnosis of the patients. Bilateral lower extremity sural sensory responses of the patients will be taken. In the antidromic method in sural nerve conduction examination, the bipolar superficial electrode is placed behind the lateral malleolus; stimulation will be made with bipolar surface electrodes 12-15 cm proximal to the recording site. Initial latency should be <3.8 ms, amplitude > 10 Mv, and conduction velocity > 36 m/sec in the sensory response of the sural nerve.

Sural Nerve Ultrasonographic measurement:

Sural nerve ultrasonography (US) will be performed by another clinician (M.A.L) who is experienced in musculoskeletal ultrasonography and unaware of clinical evaluation, using a 6-18 Mhz linear probe (Mindray -UMT 200, United States). Both sural nerve joints of the participants will be evaluated. The participant will lie on the stretcher in the prone position, the ankle will be out of the bed. The 14 cm above the malleolus will be marked as the mainline, the nerve will be detected in the lateral of the tendon of the gastrocnemius muscle and the proximal of the saphenous vein. Nerve diameter measurement will be measured 3 times in mm2 and the average will be taken. Then, possible inflammatory pathologies will be ruled out by providing clinical confirmation using the Doppler mode.

Fibromyalgia Impact Questionnaire (FIQ). Functional status assessment will be evaluated with the Fibromyalgia Impact Questionnaire (FİQ). The validity and reliability version of the questionnaire was done by researchers. This scale measures 10 different features: physical function, well-being, not being able to go to work, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety, and depression. With the exception of the well-being trait, low scores indicate recovery or less affliction. The maximum score is 100. The average of fibromyalgia scores 50, while more severely affected, usually score above 70 is used.

Neuropathic pain questionnaire:

Its Turkish validity and reliability were established. It is a questionnaire to evaluate and treat the pain of participants with pain problems, to determine exactly what type of pain they have, whether they have changed over time and their pain is in one or more areas. It consists of 12 questions. Each question is scored between 0 and 100 points. For example; If you do not have burning pain, you can score "0". If you have the worst type of burning pain imaginable, you can rate it "100". If your pain is somewhere in-between and doesn't fit either situation, choose a number that fits your pain. For each of the 12 items, the participant's scores are noted. Graded scores are multiplied by the coefficients determined for each question. All the resulting values are summed up, including fixed numbers. The result of the sum reflects the discriminant function score. Participants with a score below 0 are predicted to have non-neuropathic pain, while those with a score of 0 or higher are predicted to have neuropathic pain.

In this study; the aim is to compare the results by evaluating the ultrasonographic and electromyographic measurements of the sural nerve between the groups and to determine the correlation of these results to each other and to the FIQ, neuropathic pain questionnaire in both groups.

ELIGIBILITY:
Inclusion Criteria:

Criteria for Inclusion in the Research:

* over 18 years old,
* Able to communicate in Turkish,
* It was planned to consist of individuals who were literate and agreed to participate in the study among patients without psychiatric disease.

Exclusion Criteria:

* Having a sensory defect or a disease that may cause sensory defect (DM, -Polyneuropathy, Parkinson's, Alzheimer's disease)
* Kby, patients with uncontrollable hormonal abnormality
* HIV, hcv, hbv, vasculitis, connective tissue disease
* Patients who have undergone saphenous vein surgery
* Patients who have received radiotherapy in the leg area
* Patients with cardiac pacemaker
* Patients undergoing treatment for malignancy and who have received kt that may lead to neuropathy
* Having problems with reading and writing,communication problem
* Those who are pregnant
* Those who are deficient in B12 and other B group vitamins

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FEA) | 12 weeks
  Functional status assessment will be evaluated with the Fibromyalgia Impact Questionnaire (FEA). The validity and reliability version of the questionnaire was done by Sarmer et al. made by (12). This scale; It measures 10 different features: physical function, well-being, not being able to go to work, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. With the exception of the well-being trait, low scores indicate recovery or less affliction. The maximum score is 100. The average FM patient scores 50, while more severely affected FM patients usually score above 70.All patients with and without fibromyalgia diagnosis who participated in the study will fill out a questionnaire, and their relationship with each other will be evaluated by making ultrasonographic and electromyographic measurement evaluations of the sural nerve. there is no follow-up planned in the future as the study participants will not be administered.

SECONDARY OUTCOMES:
Neuropathic pain questionnaire | 12 weeks
  Its Turkish validity and reliability were established. It is a questionnaire to evaluate and treat the pain of patients with pain problems, to determine exactly what type of pain they have, whether they have changed over time and their pain is in one or more areas. It consists of 12 questions. Each question is scored between 0 and 100 points. For example; If you do not have burning pain, you can score "0". If you have the worst type of burning pain imaginable, you can rate it "100".It is a questionnaire to evaluate and treat the pain of patients with pain problems, to determine exactly what type of pain they have, whether they have changed over time and their pain is in one or more areas. It consists of 12 questions. Each question is scored between 0 and 100 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)